CLINICAL TRIAL: NCT01572727
Title: A Randomized, Double-blind, Placebo Controlled, Phase II/III Study of BKM120 Plus Paclitaxel in Patients With HER2 Negative Inoperable Locally Advanced or Metastatic Breast Cancer, With or Without PI3K Pathway Activation.
Brief Title: A Study of the Experimental Drug BKM120 With Paclitaxel in Patients With HER2 Negative, Locally Advanced or Metastatic Breast Cancer, With or Without PI3K Activation
Acronym: BELLE-4
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBKM120F2202; 2011-005932-24 (EudraCT Number)
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Results first posted 2017-01-27 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: BKM120; paclitaxel; breast cancer; metastatic; locally advanced; PI3K; PIK3CA; PTEN
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Hereditary Sensory and Autonomic Neuropathies | interventions — Paclitaxel; NVP-BKM120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BKM120 and paclitaxel (Experimental): Adult females with histologically confirmed, inoperable, locally advanced or metastatic HER2- BC who received study drug plus paclitaxel.
  Interventions: Drug: Paclitaxel; Drug: BKM120
- Placebo and paclitaxel (Active Comparator): Adult females with histologically confirmed, inoperable, locally advanced or metastatic HER2- BC who received placebo plus paclitaxel.
  Interventions: Drug: Paclitaxel; Drug: BKM120 matching placebo

INTERVENTIONS:
Drug: Paclitaxel — intravenous paclitaxel 80 mg/m2 per week given until progression
  Other Names: Taxol
Drug: BKM120 matching placebo — Buparlisib maching plaxcebo were supplied as 100 mg and 50 mg hard gelatin capsules.
  Buparlisib placebo was dosed on a flat scale of mg/day and was not adjusted to body weight or body surface area.
  Arms: Placebo and paclitaxel
Drug: BKM120 — Buparlisib (BKM120) were supplied as 100 mg and 50 mg hard gelatin capsules. Buparlisib was dosed on a flat scale of mg/day and was not adjusted to body weight or body surface area.
  Other Names: Buparlisib
  Arms: BKM120 and paclitaxel

SUMMARY:
This study evaluated whether the addition of daily BKM120 to weekly paclitaxel was effective and safe in treating patients with HER2- locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
Based on the efficacy results at the time of the interim analyses, the DMC recommended stopping the study at Phase II during the interim as it met the protocol pre-specified futility criteria. Consequently, the Phase III portion of the study was not conducted.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer that is locally advanced or metastatic
* HER2 negative disease, and a known hormone receptor status - ER/PgR (common breast cancer classification tests)
* A tumor sample must be shipped to a central lab for identification of biomarkers (PI3K activation status) before randomization
* Adequate bone marrow and organ function
* Measurable or non-measurable disease

Exclusion Criteria:

* Prior chemotherapy for locally advanced or metastatic disease
* Previous treatment with PI3K or AKT inhibitors
* Patient has symptomatic CNS metastases
* Concurrent malignancy or malignancy within 3 years of study enrollment
* Hematopoietic colony-stimulating growth factors or radiation within 2-4 weeks prior to starting study drug
* Increasing or chronic treatment (> 5 days) with corticosteroids or another immunosuppressive agent
* Active heart (cardiac) disease as defined in the protocol
* Known hypersensitivity or contraindications to use paclitaxel
* Pregnant or nursing (lactating) woman
* Certain scores on an anxiety and depression mood questionaire given at screening
* Other protocol defined criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (101):
- United States (21):
  - Ironwood Cancer and Research Centers SC, Chandler, Arizona
  - Arizona Oncology Associates Dept of Oncology, Phoenix, Arizona
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - California Cancer Care Marian Speciality, Greenbrae, California
  - Rocky Mountain Cancer Centers RMCC Hale Pkwy, Greenwood Village, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute SC, Tampa, Florida
  - Emory University School of Medicine/Winship Cancer Institute Dept.of WinshipCancerInst. (2), Atlanta, Georgia
  - Northwest Georgia Oncology Center NW Georgia Onc, Marietta, Georgia
  - University of Kansas Cancer Center Univ Kansas 2, Kansas City, Kansas
  - Norton Healthcare, Inc., Louisville, Kentucky
  - Washington University School of Medicine Regulatory, St Louis, Missouri
  - University of Nebraska Medical Center Unv Nebraska Med Ctr (2), Omaha, Nebraska
  - University of New Mexico Cancer Research Center Dept of Univ New Mexico, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C. Dept. of New York Oncology. PC, Troy, New York
  - Ohio State Comprehensive Cancer Center/James Cancer Hospital SC-1, Columbus, Ohio
  - University of Oklahoma Health Sciences Center OUHSC 2, Oklahoma City, Oklahoma
  - Northwest Cancer Specialists Vancouver Loc, Portland, Oregon
  - Baylor Health Care System/Sammons Cancer Center Baylor Texas Oncology, Dallas, Texas
  - University of Texas Southwestern Medical Center Harry Hines, Dallas, Texas
  - Cancer Care Centers of South Texas / HOAST CCC of So. TX- San Antonio, San Antonio, Texas
  - Medical Oncology & Hematology Associates of Northern VA Med Onc Hem Northern VA, Reston, Virginia
- Australia (4):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Geelong, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (5):
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Ottignies
  - Novartis Investigative Site, Sint-Niklaas
  - Novartis Investigative Site, Wilrijk
- Brazil (2):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Montreal, Quebec, Canada
- Czechia (3):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- France (10):
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Saint-Herblain
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Germany (9):
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Ravensburg
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Hong Kong SAR, Hong Kong
- Hungary (3):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Szolnok
- Israel (2):
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
- Japan (9):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Koto, Tokyo
- Netherlands (2):
  - Novartis Investigative Site, Breda, Netherlands
  - Novartis Investigative Site, Rotterdam
- Russia (2):
  - Novartis Investigative Site, Saint Petersburg, Russia
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Novartis Investigative Site, Johannesburg, South Africa
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (10):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz de Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Zaragoza, Zaragoza
- Taiwan (3):
  - Novartis Investigative Site, Taipei, Taiwan
  - Novartis Investigative Site, Kuei-Shan Chiang, Taoyuan/ Taiwan ROC
  - Novartis Investigative Site, New Taipei City
- United Kingdom (4):
  - Novartis Investigative Site, Maidstone, Kent
  - Novartis Investigative Site, Glasgow - Scotland
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Metropolitan Borough of Wirral

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 416 patients randomized patients, 405 received the study treatment & 403 had at least 1 post-baseline safety assessment. Randomization of patients was stopped following DMC decision & all but 5 still benefiting from the treatment were discontinued. The DMC decision was based on pre-defined futility criteria at time of the adaptive interim analysis.
Pre-assignment Details: A total of approximately 524 patients were to be randomized in a 1:1 ratio to one of the two treatment arms irrespective of the adaptation decision to continue in the full or PI3K pathway activated subpopulation. Randomization was stratified by PI3K activation and Hormone Receptor status.
Period: Overall Study
Arm/Group | BKM120 and Paclitaxel | Placebo and Paclitaxel
Started | 207 | 209
Pts With Treatment + Safety Assessment | 202 (patients who received study treatment and had at least one post-baseline safety assessment) | 201 (patients who received study treatment and had at least one post-baseline safety assessment)
Completed | 0 | 0
Not Completed | 207 | 209
Not completed — Adverse Event | 43 | 15
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 23 | 9
Not completed — Progressive disease | 59 | 82
Not completed — Protocol Violation | 0 | 1
Not completed — Study terminated by sponsor | 61 | 83
Not completed — Parent/guardian decision | 14 | 9
Not completed — Death | 2 | 2
Not completed — Untreated | 4 | 7

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all patients who were randomized to study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BKM120 and Paclitaxel | Placebo and Paclitaxel | Total
Number analyzed (Participants) | 207 | 209 | 416
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.1 (11.13) | 55.6 (10.48) | 54.9 (10.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207 | 209 | 416
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)Assessed by Local Investigator's Assessment (Phase ll)
Description: PFS was defined as the time from the date of randomization to the date of the event, defined as the first radiologically documented disease progression or death due to any cause. Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Every 8 weeks from randomization until disease progression up to 10 months after futility was analyzed
Population: FAS per Expert Report: All pts randomized to study treatment. Per ITT principle, pts were analyzed according to treatment & strata. FAS was primary population for analysis of efficacy endpoints at interim. 338 pts were randomized (between 16-Aug-2012 & 07-Jun-2014) in 1:1 ratio to buparlisib + paclitaxel arm N=168 or placebo + paclitaxel arm N=170.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 168 | 170
Months | 8.0 [7.2 to 9.2] | 9.2 [7.3 to 11.0]
Statistical Analysis 1: Comparison: BKM120 and Paclitaxel vs Placebo and Paclitaxel; Test type: Superiority or Other; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.82 to 1.68]

2. Secondary Outcome: Overall Survival by Kaplan-Meier Estimate (Phase ll)
Description: Overall survival (OS) was defined as the time from date of randomization to date of death due to any cause. If a patient was not known to have died by the date of analysis cut-off, OS was censored at the date of last contact.
Time Frame: every 3 months until death, lost to follow-up, or withdrawal of consent to survival follow-up, up to 10 months after futility was analyzed
Population: Full analysis set (FAS) comprises all patients who were randomized to study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BKM120 and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 207 | 209
Months | 29.5 [25.0 to 30.0] | NA [NA to NA] — N/A = Given the fact that patients were discontinued after the interim analysis the number of participants with events was too low to analyze.

3. Secondary Outcome: Overall Response Rate (Phase ll)
Description: Percentage of patients with best overall response of complete response (CR) or partial response (PR) based on local investigator's assessment according to RECIST v1.1. According to this criteria, CR = at least two determinations of CR at least 4 weeks apart before progression; PR = at least two determinations of PR or better at least 4 weeks apart before progression (and not qualifying for a CR). Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: every 8 weeks after randomization Up to 3 months after end of Treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BKM120 and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 168 | 170
Percentage of participants | 22.6 [16.5 to 29.7] | 27.1 [20.5 to 34.4]

4. Secondary Outcome: Duration of Response (Phase Lll)
Description: time from the date of the first documented response (CR or PR, which had to be confirmed subsequently) to the date of the first radiologically documented disease progression or death due to disease
Time Frame: every 8 weeks after randomization Up to 3 months after end of Treatment
Population: PFS, ORR and CBR were analyzed and reported at the interim analysis. Given the study met the futility analysis per protocol, the duration of response was removed as a secondary endpoint in the final analysis and consequently not analyzed.
Arm/Group | BKM120 and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Response (Phase Lll)
Description: time from date of randomization until first documented response (CR or PR, which has to be confirmed subsequently).
Time Frame: every 8 weeks after randomization Up to 3 months after end of Treatment
Population: PFS, ORR and CBR were analyzed and reported at the interim analysis. Given the study met the futility analysis per protocol, time to response was removed as a secondary endpoint in the final analysis and consequently not analyzed.
Arm/Group | BKM120 and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Clinical Benefit Rate (CBR) (Phase ll)
Description: CBR was defined as the percentage of patients with an overall response of CR or PR or SD or non-CR/non-PD lasting more than 24 weeks based on local Investigator's assessment according to RECIST v1.1.
Time Frame: every 8 weeks after randomization Up to 3 months after end of Treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BKM120 and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 168 | 170
Percentage of participants | 26.2 [19.7 to 33.5] | 32.9 [25.9 to 40.6]

7. Secondary Outcome: Plasma Concentration-time Profiles of BKM120 - Pharmacokinetics (PK) (Phase Lll)
Description: Summary statistics for PK: plasma concentration-time profiles of BKM120 and appropriate individual PK parameters based on population PK model , if deemed appropriate; each cycle = 28 days
Time Frame: Cycle 1 day 1, 15, 16, 22 and Cycle 2 day 1.
Population: PFS, ORR and CBR were analyzed and reported at the interim analysis. Given the study met the futility analysis per protocol, the plasma concentration-time profiles was removed as a secondary endpoint in the final analysis and consequently not analyzed.
Arm/Group | BKM120 and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Time to Definitive Deterioration of ECOG Performance Status (Phase Lll)
Description: Time to definitive deterioration of the ECOG performance status from baseline
Time Frame: every 4 weeks
Population: PFS, ORR and CBR were analyzed and reported at the interim analysis. Given the study met the futility analysis per protocol, the time to definitive deterioration of ECOG performance status was removed as a secondary endpoint in the final analysis and consequently not analyzed.
Arm/Group | BKM120 and Paclitaxel | Placebo and Paclitaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Among 416 randomized patients, 405 patients received the study treatment. Of them, 403 patients had at least one post-baseline safety assessment.
Groups:
- Buparlisib (BKM120) 100 mg Plus Paclitaxel 80 mg Per m2: Adult females with histologically confirmed, inoperable, locally advanced or metastatic HER2- BC who received study drug plus paclitaxel
- Placebo 100 mg Plus Paclitaxel 80 mg Per m2: Adult females with histologically confirmed, inoperable, locally advanced or metastatic HER2- BC who received placebo plus paclitaxel
Arm/Group | Buparlisib (BKM120) 100 mg Plus Paclitaxel 80 mg Per m2 | Placebo 100 mg Plus Paclitaxel 80 mg Per m2
Serious Adverse Events (participants affected / at risk) | 61/202 | 42/201
Other Adverse Events (participants affected / at risk) | 196/202 | 188/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Buparlisib (BKM120) 100 mg Plus Paclitaxel 80 mg Per m2 (N=202) | Placebo 100 mg Plus Paclitaxel 80 mg Per m2 (N=201)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
CATARACT (Eye disorders) | 1 | 1
OPTIC NEUROPATHY (Eye disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 5 | 3
NAUSEA (Gastrointestinal disorders) | 1 | 1
PANCREATITIS (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 2 | 1
ASTHENIA (General disorders) | 3 | 0
FACE OEDEMA (General disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 3
LOCALISED OEDEMA (General disorders) | 1 | 0
MALAISE (General disorders) | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 1
PYREXIA (General disorders) | 7 | 3
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 0 | 1
HYPERSENSITIVITY (Immune system disorders) | 1 | 1
ABSCESS LIMB (Infections and infestations) | 0 | 1
CELLULITIS (Infections and infestations) | 1 | 5
DEVICE RELATED INFECTION (Infections and infestations) | 2 | 2
GASTROENTERITIS (Infections and infestations) | 0 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 0 | 1
INFUSION SITE INFECTION (Infections and infestations) | 1 | 0
MENINGITIS (Infections and infestations) | 0 | 1
PNEUMOCYSTIS JIROVECII INFECTION (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
PYELONEPHRITIS (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 3 | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 4 | 1
FALL (Injury, poisoning and procedural complications) | 2 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 1 | 0
POST-TRAUMATIC PAIN (Injury, poisoning and procedural complications) | 1 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
EJECTION FRACTION DECREASED (Investigations) | 1 | 0
LYMPHOCYTE COUNT INCREASED (Investigations) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 3
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 1
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
BRACHIAL PLEXOPATHY (Nervous system disorders) | 1 | 0
BRAIN COMPRESSION (Nervous system disorders) | 0 | 1
BRAIN OEDEMA (Nervous system disorders) | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 1
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
HEMIPARESIS (Nervous system disorders) | 1 | 0
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0
SEIZURE (Nervous system disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 2
ACUTE PSYCHOSIS (Psychiatric disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 2 | 1
DELIRIUM (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0
MENTAL DISORDER (Psychiatric disorders) | 2 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 2 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
BREAST HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
BREAST ULCERATION (Reproductive system and breast disorders) | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 6 | 1
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RASH (Skin and subcutaneous tissue disorders) | 2 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN MASS (Skin and subcutaneous tissue disorders) | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2 | 0
SWELLING FACE (Skin and subcutaneous tissue disorders) | 1 | 0
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 1 | 0
DIET NONCOMPLIANCE (Social circumstances) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 3 | 1
HYPERTENSION (Vascular disorders) | 2 | 0
VENA CAVA THROMBOSIS (Vascular disorders) | 1 | 0
VENOUS THROMBOSIS (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Buparlisib (BKM120) 100 mg Plus Paclitaxel 80 mg Per m2 (N=202) | Placebo 100 mg Plus Paclitaxel 80 mg Per m2 (N=201)
ANAEMIA (Blood and lymphatic system disorders) | 46 | 51
NEUTROPENIA (Blood and lymphatic system disorders) | 64 | 54
LACRIMATION INCREASED (Eye disorders) | 12 | 17
VISION BLURRED (Eye disorders) | 19 | 7
ABDOMINAL PAIN (Gastrointestinal disorders) | 27 | 22
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 11 | 14
CONSTIPATION (Gastrointestinal disorders) | 47 | 38
DIARRHOEA (Gastrointestinal disorders) | 109 | 68
DRY MOUTH (Gastrointestinal disorders) | 12 | 10
DYSPEPSIA (Gastrointestinal disorders) | 23 | 15
NAUSEA (Gastrointestinal disorders) | 83 | 51
STOMATITIS (Gastrointestinal disorders) | 56 | 24
VOMITING (Gastrointestinal disorders) | 39 | 30
ASTHENIA (General disorders) | 48 | 45
FATIGUE (General disorders) | 67 | 64
NON-CARDIAC CHEST PAIN (General disorders) | 4 | 11
OEDEMA PERIPHERAL (General disorders) | 21 | 50
PAIN (General disorders) | 9 | 11
PYREXIA (General disorders) | 29 | 19
RHINITIS (Infections and infestations) | 11 | 9
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 23
URINARY TRACT INFECTION (Infections and infestations) | 18 | 18
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 35 | 12
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 30 | 11
BLOOD GLUCOSE INCREASED (Investigations) | 13 | 10
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 7 | 12
NEUTROPHIL COUNT DECREASED (Investigations) | 15 | 15
WEIGHT DECREASED (Investigations) | 30 | 14
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 10 | 14
DECREASED APPETITE (Metabolism and nutrition disorders) | 64 | 26
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 82 | 22
HYPOKALAEMIA (Metabolism and nutrition disorders) | 19 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 23 | 32
BACK PAIN (Musculoskeletal and connective tissue disorders) | 21 | 22
BONE PAIN (Musculoskeletal and connective tissue disorders) | 10 | 14
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 8 | 12
MYALGIA (Musculoskeletal and connective tissue disorders) | 22 | 27
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 27 | 40
DIZZINESS (Nervous system disorders) | 33 | 21
DYSGEUSIA (Nervous system disorders) | 39 | 34
HEADACHE (Nervous system disorders) | 35 | 37
NEUROPATHY PERIPHERAL (Nervous system disorders) | 50 | 48
PARAESTHESIA (Nervous system disorders) | 25 | 34
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 31 | 31
ANXIETY (Psychiatric disorders) | 41 | 31
DEPRESSION (Psychiatric disorders) | 50 | 17
INSOMNIA (Psychiatric disorders) | 31 | 33
MOOD ALTERED (Psychiatric disorders) | 11 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 40 | 28
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 26 | 21
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 29 | 33
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 12 | 16
ALOPECIA (Skin and subcutaneous tissue disorders) | 103 | 104
DRY SKIN (Skin and subcutaneous tissue disorders) | 28 | 13
ERYTHEMA (Skin and subcutaneous tissue disorders) | 11 | 17
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 7 | 14
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 7 | 19
ONYCHOMADESIS (Skin and subcutaneous tissue disorders) | 7 | 11
PRURITUS (Skin and subcutaneous tissue disorders) | 32 | 30
RASH (Skin and subcutaneous tissue disorders) | 86 | 43
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 12 | 8
FLUSHING (Vascular disorders) | 7 | 11
HYPERTENSION (Vascular disorders) | 17 | 10
LYMPHOEDEMA (Vascular disorders) | 7 | 16

LIMITATIONS AND CAVEATS:
Safety set: all randomized pts who received at least 1 dose of the study treatment (either buparlisib + paclitaxel or matching placebo + paclitaxel) & had at least 1 post-baseline safety assessment;13 of 416 pts didn't meet this criteria; safety =403

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.